CLINICAL TRIAL: NCT02366481
Title: Vitamin K and Glucose Metabolism in Adults at Risk for Diabetes
Brief Title: Vitamin K and Glucose Metabolism in Adults at Risk for Diabetes (Vita-K 'n' Adults Study)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Augusta University (Other)
Collaborators: University of Alabama at Birmingham (Other); Yale University (Other); Tufts University (Other)
Responsible Party: Principal Investigator, Norman Pollock, Associate Professor, Department of Medicine, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 620511; 16GRNT31090037 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2015-02-12; First posted 2015-02-19 (Estimated); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Obesity; Insulin Resistance; Insulin Sensitivity; Beta-Cell Dysfunction; Prediabetes
Keywords: Vitamin K; Vitamin K2; Menaquinone-7; Osteocalcin; Adults; Obesity; Insulin resistance; Insulin sensitivity; Beta-cell function; Prediabetes
MeSH Terms: conditions — Obesity; Insulin Resistance; Prediabetic State | interventions — menaquinone 7

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo-Control (Placebo Comparator): The placebo-control group will take two placebo softgel capsules every day for 8 weeks.
  Interventions: Dietary Supplement: Placebo
- Low-Dose Vitamin K2 (90-mcg/d) (Active Comparator): The low-dose vitamin K group will take one 90-mcg vitamin K2 (menaquinone-7) softgel capsule and one placebo softgel capsule every day for 8 weeks.
  Interventions: Dietary Supplement: Low-Dose Vitamin K2 Supplement (menaquinone-7; 90-mcg/d)
- High-Dose Vitamin K2 (180-mcg/d) (Active Comparator): The high-dose vitamin K group will take two 90-mcg vitamin K2 (menaquinone-7) softgel capsules every day for 8 weeks.
  Interventions: Dietary Supplement: High-Dose Vitamin K2 Supplement (menaquinone-7; 180-mcg/d)

INTERVENTIONS:
Dietary Supplement: Placebo — Two placebo softgel capsules (containing no vitamin K2) every day for 8 weeks.
  Arms: Placebo-Control
Dietary Supplement: Low-Dose Vitamin K2 Supplement (menaquinone-7; 90-mcg/d) — One 90-mcg vitamin K2 softgel capsules (containing no vitamin K2) and one placebo softgel capsule everyday for 8 weeks.
  Arms: Low-Dose Vitamin K2 (90-mcg/d)
Dietary Supplement: High-Dose Vitamin K2 Supplement (menaquinone-7; 180-mcg/d) — Two 90-mcg vitamin K2 softgel capsules every day for 8 weeks.
  Arms: High-Dose Vitamin K2 (180-mcg/d)

SUMMARY:
Given that glutamate carboxylation or decarboxylation is key to the metabolic role of osteocalcin (at least in mouse models) and that carboxylation is vitamin K dependent, it is critical to isolate the effect of vitamin K manipulation on carboxylation of osteocalcin and its subsequent effect on glucose metabolism in clinical trials. The purpose of this randomized, double-blind, placebo-controlled clinical trial in adults is to determine whether eight weeks of daily supplementation with vitamin K2 (menaquinone-7) can improve markers in blood associated with diabetes risk.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults between 18 and 65 years old
2. Subject understands the study protocol and agrees to comply with it
3. Informed Consent Form signed by the subject

Exclusion Criteria:

1. Subjects using vitamin supplements containing vitamin k
2. Subjects with (a history of) metabolic or gastrointestinal diseases including hepatic disorders
3. Subjects presenting chronic degenerative and/or inflammatory diseases
4. Subjects receiving systemic treatment or topical treatment likely to interfere with evaluation of the study parameters (salicylates, antibiotics)
5. Subjects receiving corticosteroid treatment
6. Subjects using oral anticoagulants
7. Subjects with a history of soy allergy
8. Subjects who have participated in a clinical study more recently than one month before the current study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-02; Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in insulin sensitivity | Change from baseline in insulin sensitivity at 8 weeks
  Insulin sensitivity will be calculated from plasma insulin and glucose concentrations measured during a 2-hour oral glucose tolerance test by using the oral glucose minimal model.
Change in beta-cell function | Change from baseline in beta-cell function at 8 weeks
  Beta-cell function, as assessed by dynamic beta-cell responsitivity, will be calculated from plasma glucose and C-peptide concentrations measured during a 2-hour oral glucose tolerance test by using the oral C-peptide minimal model.

SECONDARY OUTCOMES:
Change in prothrombin time (PT) | Change from baseline in PT at 8 weeks
Change in activated partial thromboplastin time (aPTT) | Change from baseline in aPTT at 8 weeks
Change in arterial stiffness (PWV) | Change from baseline in arterial stiffness at 8 weeks
  Arterial stiffness will be assessed using carotid-femoral pulse wave velocity (PWV) by applanation tonometry.
Change in endothelial function (FMD) | Change from baseline in endothelial function at 8 weeks
  Endothelial function will be assessed using brachial artery flow-mediated dilation (FMD) by ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Norman K Pollock, Ph.D., Principal Investigator — Department of Pediatrics, Medical College of Georgia, Augusta University
Locations (1):
- Medical College of Georgia; Augusta University, Augusta, Georgia, United States

REFERENCES:
- [Background] Pollock NK, Bernard PJ, Gower BA, Gundberg CM, Wenger K, Misra S, Bassali RW, Davis CL. Lower uncarboxylated osteocalcin concentrations in children with prediabetes is associated with beta-cell function. J Clin Endocrinol Metab. 2011 Jul;96(7):E1092-9. doi: 10.1210/jc.2010-2731. Epub 2011 Apr 20. PMID 21508147
- [Background] Gower BA, Pollock NK, Casazza K, Clemens TL, Goree LL, Granger WM. Associations of total and undercarboxylated osteocalcin with peripheral and hepatic insulin sensitivity and beta-cell function in overweight adults. J Clin Endocrinol Metab. 2013 Jul;98(7):E1173-80. doi: 10.1210/jc.2013-1203. Epub 2013 Apr 24. PMID 23616149
- [Background] Booth SL, Centi A, Smith SR, Gundberg C. The role of osteocalcin in human glucose metabolism: marker or mediator? Nat Rev Endocrinol. 2013 Jan;9(1):43-55. doi: 10.1038/nrendo.2012.201. Epub 2012 Nov 13. PMID 23147574
- [Background] Pollock NK. Childhood obesity, bone development, and cardiometabolic risk factors. Mol Cell Endocrinol. 2015 Jul 15;410:52-63. doi: 10.1016/j.mce.2015.03.016. Epub 2015 Mar 27. PMID 25817542